CLINICAL TRIAL: NCT06100406
Title: Sound Healing for Anxiety: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Consciousness and Healing Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT001
Record Dates: First submitted 2023-10-16; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Anxiety; Mental Health Issue; Anxiety Generalized; Anxiety State
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Intervention versus waitlist control. The control group will have the option to receive the intervention after the study is completed.
Who Masked: Outcomes Assessor
Masking Description: Once randomized, the participants will know they are receiving the intervention. Outcomes assessor will be masked for data analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Biofield Tuning is a non-invasive, non-medical therapeutic practice in which a resonating tuning fork is used to identify and re-balance off-the-body sites at which perturbations in the tuning fork sound are detected. The description of the intervention has been provided by Biofield Tuning Practitioners and thus describes the practitioner's experience and process while performing the intervention.
  For this study, the Biofield Tuning practitioner will be using a "hologram" of the participant's body since the intervention will be performed remotely. A "hologram" is when a BT practitioner imagines the body of the participant on the table in front of them. This approach was used successfully for our last feasibility study suggesting an impact of the virtually delivered BT intervention on anxiety.
  Interventions: Other: Biofield tuning
- Waitlist control (No Intervention): The waitlist control group will complete the same weekly self-report questionnaires outlined in the protocol as the intervention group and weekly audio recordings. Following their one-month follow-up questionnaire, those in the waitlist group will be offered a BT session at no cost.

INTERVENTIONS:
Other: Biofield tuning — Biofield Tuning is a non-invasive, non-medical therapeutic practice in which a resonating tuning fork is used to identify and re-balance off-the-body sites at which perturbations in the tuning fork sound are detected.
  Other Names: sound healing
  Arms: Intervention

SUMMARY:
The goal of this randomized controlled trial is to compare a novel sound healing approach, biofield tuning, to a waitlist control group in a healthy adult population naive to the intervention. The main questions it aims to answer are:

* Is there a significant reduction in state and trait anxiety as measured by the State-Trait Anxiety Index (STAI) with biofield tuning compared to waitlist control?
* Are there significant reductions in negative affect, as well as increases in self-compassion, positive affect, and interoceptive awareness in the intervention group?
* What are the relationships between changes in anxiety symptoms, negative affect words, and microbiome changes in participants who have undergone this biofield intervention?

Participants will be:

* Randomized to intervention/control
* Recieve 5 sound healing interventions weekly
* Asked to complete surveys and audio prompts throughout the intervention
* Asked to provide a microbiome sample pre- and post-intervention

DETAILED DESCRIPTION:
There is an increasing rate of anxiety among the US population, without adequate amounts of resources for treatment. Current pharmacological and psychological treatments for generalized anxiety disorder delivered by doctors, nurses, and clinical psychologists are often expensive and not freely available for many who need effective interventions for anxiety. A novel sound healing approach, Biofield Tuning (BT), has suggested potential benefits to those suffering from generalized anxiety. This intervention, while requiring training and certification, allows for holistic health practitioners to treat anxiety as a complementary mind-body therapy for those seeking relief for anxiety.

Intervention. BT is a non-invasive, non-medical therapeutic practice developed by Eileen Day McKusick. BT Practitioners use a tuning fork to identify off-the-body sites at which perturbations in the tuning fork sound are detected. Such sites are described by BT practitioners as storing health-related information within the human biofield. Practitioners describe the process of BT as assessing and clearing perturbations in the human biofield to foster healing.

Previous Feasibility Study. Our initial cohort study showed that conducting research for this novel sound healing approach online was feasible and suggested clinical benefits for people struggling with moderate to severe generalized anxiety, as noted in our peer-reviewed scientific publication. This RCT is designed to build upon the previous cohort study by comparing this intervention with a control group to further determine the effectiveness of BT compared to treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older (≥ 18)
* Biofield-tuning naive (have never had a session of biofield tuning before)
* Speak and understand English at a native level
* Have a score ≥10 on the Generalized Anxiety Disorder 7-item (GAD-7) scale
* Have regular access to a computer
* Have experience using a computer
* Be comfortable using Zoom and completing data collection activities online and over the phone

Exclusion Criteria:

* Suffering from any severe psychological, physical, or cognitive disease or impairment.
* An active diagnosis or history of suicidality, Post-Traumatic Stress Disorder (PTSD), schizophrenia, or psychotic disorders. This includes history or current suicidality, suicide ideation, and intent to harm self or others.
* Women who are pregnant or nursing.
* Having an electronically implanted device, excluding cochlear implants.
* Currently seeking treatment for an active cancer.
* Currently has an untreated serious illness (e.g. heart disease, diabetes, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks
  The main objective is to assess whether virtually-delivered biofield tuning can significantly reduce moderate to high levels of generalized anxiety as measured by the State Trait Anxiety Index (STAI).

SECONDARY OUTCOMES:
Anxiety 1-month | 1-month post-intervention
  We also aim to understand how long BT intervention effects may last with a 1-month follow up as measured by the STAI.
Positive and Negative Affect | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 1-month post-intervention
  as measured by the Positive and Negative Affect Scale-Short Form (PANAS)
Interoceptive awareness | Baseline, at 5 weeks
  as measured by the Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2)
mental health recovery | Baseline, at 3 weeks, 5 weeks and 1-month post-intervention
  as measured by the Recovery Assessment Scale- Revised (RAS-r). Scores range from 24 to 120. Items are rated from 1 to 5. Higher scores indicate higher levels of recovery.
stress | Baseline, at 3 weeks, 5 weeks and 1-month post-intervention
  as measured by the Perceived Stress Scale (PSS). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
self compassion | Baseline, at 3 weeks, 5 weeks and 1-month post-intervention
  as measured by the Self-Compassion Scale-Short Form (SCS-SF). The total score is an overall indication of self-compassion, with a higher score indicating more self-compassion.
perceived social support | Baseline, at 3 weeks, 5 weeks and 1-month post-intervention
  as measured by the Multidimensional Scale of Perceived Social Support (MSPSS)
relationship with practitioner | at 1 week, 3 weeks, and 5 weeks
  as measured by a Practitioner Relationship questionnaire
depressive symptoms | Baseline, at 3 weeks, 5 weeks and 1-month post-intervention
  as measured by the PHQ-9

OTHER OUTCOMES:
Spoken Language | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 1-month post-intervention
  As measured by a spoken prompt that will be recorded
Microbiome changes | Baseline and 5 weeks
  as measured by a microbiome sample

CONTACTS AND LOCATIONS:
Overall Officials: Shamini Jain, PhD, Principal Investigator — Consciousness and Healing Initiative; Hemal H Patel, PhD, Principal Investigator — University of California, San Diego; Cassandra Vieten, PhD, Principal Investigator — University of California, San Diego

IPD SHARING:
Plan to Share IPD: Yes
No individual data or identifiers will be shared with other researchers.
Supporting Information: Analytic Code
Time Frame: 2 years
Access Criteria: Subject code blinded. Treatment code blinded and unblinded for analyses.

REFERENCES:
- [Background] Jain S, Hammerschlag R, Mills P, Cohen L, Krieger R, Vieten C, Lutgendorf S. Clinical Studies of Biofield Therapies: Summary, Methodological Challenges, and Recommendations. Glob Adv Health Med. 2015 Nov;4(Suppl):58-66. doi: 10.7453/gahmj.2015.034.suppl. Epub 2015 Nov 1. PMID 26665043
- [Result] Jain S, McKusick E, Ciccone L, Sprengel M, Ritenbaugh C. Sound healing reduces generalized anxiety during the pandemic: A feasibility study. Complement Ther Med. 2023 Jun;74:102947. doi: 10.1016/j.ctim.2023.102947. Epub 2023 Apr 5. PMID 37023932